CLINICAL TRIAL: NCT06982378
Title: Effect of Glucagon-like Peptide -1 Receptor Agonist on Liver Tissue and Plasma Lipids in MASLD
Brief Title: GLP-1 RA on Liver OMICS in MASLD
Acronym: OMICS in MASLD
Status: Not yet recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Achuthan Sourianarayanane, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO00050604
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: NAFLD; Diabetes; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver tissue and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without GLP-1 RA treatment: Patients with MASLD and obesity/diabetes - on standard of care treatment but not on any GLP-1 RA
- Had GLP-1 RA treatment: Patients with MASLD and obesity/diabetes - on GLP-1 RA as a standard of care treatment
  Interventions: Drug: GLP-1 receptor agonist

INTERVENTIONS:
Drug: GLP-1 receptor agonist — on and not on treatment
  Groups: Had GLP-1 RA treatment

SUMMARY:
In patients with type II diabetes mellitus (T2DM) and obesity, an excess plasma-free fatty acid is found with an associated increased lipid accumulation in adipocytes and liver tissue. Lipid droplet accumulation in the hepatocytes is an initial step in the development of metabolic dysfunction associated steatotic liver disease (MASLD. Insulin resistance, which is associated with T2DM, mediates the inflammation of these lipids, resulting in the progression of MASLD to metabolic dysfunction associated steatotic hepatitis (MASH). Hence, in T2DM, obesity, and MASLD, changes in the lipid profile occur, and they are interrelated.

In this study, we aim to assess improvement in the lipidomic, its associated metabolic changes and evaluate the co-regulated genes in the liver tissue among patients with MASLD with intervention with GLP-1 RA, which has shown to benefit T2DM and obesity.

DETAILED DESCRIPTION:
The study involves patients with a diagnosis of MASLD by histology and have diabetes/obesity. The 'omics' ( lipidomics, proteomics, metabolites, and inflammatory profiles and transcriptomics) data of liver tissue and plasma of patients will be compared between patients who have received 1 year of GLP-1 treatment with those who did not have GLP-1 agents.

The study will evaluate the changes in different 'omics' and metabolites in the liver tissue following the use of GLP-1 agents in these patients

ELIGIBILITY:
Inclusion Criteria:

* known diagnosis of MASLD by histology, also have diabetes/ obesity
* on treatment with GLP-1 RA at stable dose

Exclusion Criteria:

* unable to have a liver biopsy, recent change in medication for diabetes or hyperlipidemia
* on immunosuppression, liver or kidney transplant
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: known diagnosis of MASLD by histology, also have diabetes/ obesity
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Changes in lipidomics profile on use of GLP-1 RA | 1 year
  Lipidomic profile being evaluated

SECONDARY OUTCOMES:
Changes in associated proteomics and transcriptomics with the use of GLP-1 RA | 1 year
  proteomic and transcriptomics profiles evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No